CLINICAL TRIAL: NCT00849563
Title: Effect of Type 2 Diabetes Genetic Risk Information on Health Behaviors and Outcomes
Acronym: TDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: deCODE genetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00011592
Record Dates: First submitted 2009-02-22; First posted 2009-02-24 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: predictive genomics; personalized medicine; personal genomics; genetic knowledge; genetic attitudes; prevention; health outcomes; behavioral
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- SRA+genetic test (Active Comparator): patients randomized to receive genetic test for type 2 diabetes risk will be followed and surveyed and will be counseled based on SAR and genetic risk for type 2 diabetes
  Interventions: Other: Standardized Risk Assessment
- SRA only (No Intervention): Patients randomized to not get genetic testing will be followed and surveyed and will be counseled based on SRA only
- no testing control (No Intervention): Patients not interested in genetic testing will be followed and surveyed. Counseling will be based on SRA only

INTERVENTIONS:
Other: Standardized Risk Assessment — patients interested in genetic testing will be randomly assigned to either get testing for type 2 diabetes or not. All arms with receive standardized risk asessements. This study is evaluating behavior after receipt of genetic risk information and different types of counseling.
  Arms: SRA+genetic test

SUMMARY:
The primary objective of the study is to assess the clinical utility of a genetic test for Type 2 diabetes risk in combination with standardized risk assessment compared with standardized risk assessment alone, and to measure whether changes in perceived risk following genetic testing for Type 2 diabetes risk are correlated with behavior change and increased concern about risk for Type 2 diabetes.

DETAILED DESCRIPTION:
One thousand outpatients will be enrolled over two years at two university-affiliated primary care clinics. Patients will be assigned to one of three study arms: those who want genetic testing for diabetes risk will be randomly assigned to either receive the testing in addition to the SRA (SRA+G) or to receive the SRA only (SRA-only). Those who do not wish to have genetic testing will receive the SRA only. All patients will be surveyed at baseline, immediately after going through the SRA (risk-counseling visit; 2-4 weeks after initial visit), at 3 months post risk counseling visit and at 12 months post risk counseling visit. BMI, waist circumference, fasting plasma glucose and insulin will be measured at baseline and 12 months. Surveys will allow us to track patients' emotional responses to diabetes risk information and changing perceptions of personal risk for Type 2 diabetes over time, and to see if these correlate with subsequent diet and exercise behaviors.

We will use a linear model to assess the effects of genetic testing among the three study groups, using HOmeostasis Model Assessment of Insulin Resistance (HOMA-IR) and weight loss as the primary outcomes. We will use generalized linear ordinal regression models to fit the ordinal survey outcomes of risk perceptions to the continuous HOMA-IR and weight outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female outpatients
* No self-reported history of diabetes
* No self-reported history of prior genetic testing for diabetes
* Not pregnant (self report)
* Are ≥18 and <81 years of age
* Scheduled to receive serum glucose test in participating clinic
* Fasting at time of blood draw (no food or drink - except water - previous 8 hours: self report)
* Able and willing to give legally effective consent
* Able and willing to participate in patient questionnaires
* Ambulatory

Exclusion Criteria:

* Previously or currently taking medications for lowering glucose (i.e., exenatide, pramlintide, metformin, rosiglitazone, pioglitazone, or future diabetes drugs) based on self-report and/or prescreening
* Self-report of current or prior diabetes diagnosis
* Self-reported prior history of genetic testing for diabetes
* Baseline serum glucose test result >125

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percentage of weight loss | 12 months

SECONDARY OUTCOMES:
Change in perceptions of personal risk for Type 2 diabetes | 12 months
Change in HOmeostasis Model Assessment of Insulin Resistance (HOMA-IR) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Ginsburg, Md, PhD, Principal Investigator — Institute for Genome Sciences and Policy, Duke University; Alex Cho, MD, Principal Investigator — Institute for Genome Sciences and Policy, Duke University; Scott Joy, MD, Principal Investigator — Duke University; Susanne Haga, PhD, Principal Investigator — Institute for Genome Sciences and Policy, Duke University; Isaac Lipkus, PhD, Principal Investigator — Institute for Genome Sciences and Policy, Duke University; Gloria Trujillo, MD, Principal Investigator — Duke University; Julianne O'Daniel, PhD, Principal Investigator — Institute for Genome Sciences and Policy, Duke University
Locations (2):
- United States (2):
  - Duke Family Medicine at Pickens, Durham, North Carolina
  - Duke Health Center at Pickett Rd, Durham, North Carolina

REFERENCES:
- [Derived] Waxler JL, O'Brien KE, Delahanty LM, Meigs JB, Florez JC, Park ER, Pober BR, Grant RW. Genetic counseling as a tool for type 2 diabetes prevention: a genetic counseling framework for common polygenetic disorders. J Genet Couns. 2012 Oct;21(5):684-91. doi: 10.1007/s10897-012-9486-x. PMID 22302620
- [Derived] Cho AH, Killeya-Jones LA, O'Daniel JM, Kawamoto K, Gallagher P, Haga S, Lucas JE, Trujillo GM, Joy SV, Ginsburg GS. Effect of genetic testing for risk of type 2 diabetes mellitus on health behaviors and outcomes: study rationale, development and design. BMC Health Serv Res. 2012 Jan 18;12:16. doi: 10.1186/1472-6963-12-16. PMID 22257365